CLINICAL TRIAL: NCT03466515
Title: Stem Cells Treatment of Complex Crohns Perianal Fistula. A Pilot Clinical Study
Brief Title: Stem Cells Treatment of Complex Crohn's Anal Fistula
Acronym: fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karam Matlub Sørensen, afdelingslæge, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S-20170140
Record Dates: First submitted 2018-03-08; First posted 2018-03-15 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Anal Fistula; Crohn Disease
Keywords: stem cells therapy
MeSH Terms: conditions — Rectal Fistula; Crohn Disease | interventions — Lipectomy

STUDY DESIGN:
Intervention Model Description: pilot study with a maximum of 20 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention (Experimental): Patients enrolled in the study will be treated for their anal fistula by surgical closure of the internal opening, debridement of the fistula and injection of patients own stem cells enriched fatty tissue around the fistula.
  Interventions: Procedure: stem cells injection

INTERVENTIONS:
Procedure: stem cells injection — two surgical interventions as day-surgery, starting with liposuction from the abdomen (about 200-300 ml), and fistula tract debridement and closure of internal opening. The external opening is excised. About 30-40 ml fresh harvested patients own fatty tissue are then injected with large needle around the fistula from internal til external opening.The resting harvested fatty tissue will be sent to stem cells (Adipose Derived Regenrative Cells ADRCs) isolation, using Cytori Celusion system®. When the stem cells isolation is completed, 4ml concentrated stem cells ( contains around 20-40 millions cells ) will be injected around the prepared fistula tract, the same site where the fresh harvested fatty tissue injected before.
  Other Names: liposuction; fistula closure

SUMMARY:
A pilot study to investigate the safety and feasibility of stem cells treatment of complex anal fistula in patients with Crohn's disease.

DETAILED DESCRIPTION:
Stem cells therapy in the management of soft tissue healing has been shown to be safe and feasible with encouraging short-term results both for crypto glandular and Crohns anal fistula. The long-term results are still insufficient but based on only a few studies conducted with small patient series and various techniques and type of stem cells. In the present study the patient's own adipose tissue derived regenerative cells (ADRCs) will be used. Traditionally the stem cells are injected into the fistula tract; however survival and retaining the stem cells in the fistula tract is problematic. Alternatively, one may apply stem cells enriched fatty tissue around and into the fistula tract. The aim of this project is to develop a method for treatment of patients with Crohns fistula. The results of conventional surgery are disappointing and followed by a high degree of recurrence and complications.

ELIGIBILITY:
Inclusion Criteria:

* patients with Crohn's anal fistulas and> 18 yrs old.

Exclusion Criteria:

* Signs of suppuration around the fistula
* Active intestinal Crohn disease not in remission
* Malignancy within 5 years
* Previous radiotherapy of the abdomen and pelvis
* BMI under 18.5
* Coagulopathy
* Fistula with side branches
* Low anal fistula
* Verified syphilis, HIV, or hepatitis on screening test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
healing | 6 months
  closure of the fistula with no secretions

SECONDARY OUTCOMES:
recurrence | 6 months
  recurrence of the fistula
time to healing | 6 months
  time required to healing of the fistula
major adverse effects | 6 months
  occurrence of infections, sepsis bleeding and allergy.
radiological healing | at 6 months
  Changes on MRI scanning
functional outcome | 6 months
  changes in Wexner incontinence score

CONTACTS AND LOCATIONS:
Overall Officials: Karam Matlub, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No